CLINICAL TRIAL: NCT05862948
Title: Accuracy of Endo-aid in Consecutive Patients Referred for Colonoscopy - ACCENDO-Colo Study
Brief Title: Accuracy of Endo-aid in Consecutive Patients Referred for Colonoscopy
Acronym: ACCENDO-Colo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Poliambulanza Istituto Ospedaliero (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: NP4834
Record Dates: First submitted 2023-05-04; First posted 2023-05-17 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Adenoma Colon; Colonic Adenoma
Keywords: ADR; CADe; Endo-AID

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CADe Colonoscopy (Experimental): Colonoscopy with the help of CADe system (ENDO-Aid)
  Interventions: Device: ENDO-Aid by Olympus
- Conventional Colonoscopy (No Intervention): Standard Colonoscopy with white light

INTERVENTIONS:
Device: ENDO-Aid by Olympus — Colonoscopy assisted by ENDO-AID device
  Arms: CADe Colonoscopy

SUMMARY:
The goal of this clinical trial is to evaluate the diagnostic yield of CADe in a consecutive population undergoing colonoscopy. The main question it aims to answer is the Adenoma Detection Rate (ADR). Participants undergoing colonoscopy will be randomized in a 1:1 ratio to either receive Computer-Aided Detection (CADe) colonoscopy or a conventional colonoscopy (CC). Researchers will compare the CADe group and the CC-group to see if CAD-e can increase the ADR significantly.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years or ≤85
* Patients undergoing screening, follow-up, or diagnostic colonoscopy

Exclusion Criteria:

* Suspected or known inflammatory bowel disease
* Colonic resection
* Taking anticoagulants or antiaggregants that contraindicate the performance of therapy
* Patients with incomplete colonoscopy
* Patients with inadequate preparation using the Boston Colonic Preparation Scale (BBPS). A cleaning quality of less than 2 points in any of the 3 colonic sections will be considered inadequate.
* Inability to provide informed consent.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1160 (Actual)
Dates: Start 2021-10-30 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Adenoma detection rate (ADR) | 1 years
  ADR defined as the proportion of patients with at least 1 adenoma detected.

SECONDARY OUTCOMES:
Polyp detection rate (PDR) | 1 years
  PDR defined as the proportion of patients with at least 1 polyp detected.
Polyp per colonoscopy (PPC) | 1 years
  PPC defined as total number of polyps resected divided by the total number of colonoscopies.
Adenoma per colonoscopy (APC) | 1 years
  APC defined as total number of histologically confirmed adenomas resected divided by the total number of colonoscopies.
Sessile serrated lesion detection rate (SSLDR) | 1 years
  SSLDR percentage of patients who have 1 or more histologically confirmed sessile serrated lesion resected divided by the total number of colonoscopies.
Advanced adenoma detection rate (AADR) | 1 years
  AADR Adenomas are classified as advanced with a size >= 10mm and/or a (tubulo)villous histology and/or high-grade dysplasia (HGD)

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Fondazione Poliambulanza, Brescia, Bs
  - Policlinico Universitario Agostino Gemelli, Roma

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Spada C, Salvi D, Ferrari C, Hassan C, Barbaro F, Belluardo N, Grazioli LM, Milluzzo SM, Olivari N, Papparella LG, Pecere S, Pesatori EV, Petruzziello L, Piccirelli S, Quadarella A, Cesaro P, Costamagna G. A comprehensive RCT in screening, surveillance, and diagnostic AI-assisted colonoscopies (ACCENDO-Colo study). Dig Liver Dis. 2025 Mar;57(3):762-769. doi: 10.1016/j.dld.2024.12.023. Epub 2025 Jan 14. PMID 39814659